CLINICAL TRIAL: NCT03701633
Title: Postpartum Uterine Artery Doppler Changes Prior and After Breastfeeding
Brief Title: Uterine Artery Doppler Changes Prior and After Breastfeeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Yaniv Zipori MD, Doctor Yaniv Zipori, Rambam Health Care Campus
Other Study IDs: 0340-17-RMB
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prior to breastfeeding - cross section: Measurements of the UtA doppler postpartum ultrasound will be carried out twice for each eligible woman on the second day postpartum. The first measurement will take place just prior to a planned breastfeeding. The second measurement will be followed immediately (within 10 min) after the breastfeeding session.
  Interventions: Diagnostic Test: Postpartum ultrasound
- After breastfeeding - cross section: Measurements of the UtA doppler postpartum ultrasound will be carried out twice for each eligible woman on the second day postpartum. The first measurement will take place just prior to a planned breastfeeding. The second measurement will be followed immediately (within 10 min) after the breastfeeding session.
  Interventions: Diagnostic Test: Postpartum ultrasound

INTERVENTIONS:
Diagnostic Test: Postpartum ultrasound — Measurements of the UtA doppler ultrasound will be carried out twice for each eligible woman on the second day postpartum. The first measurement will take place just prior to a planned breastfeeding. The second measurement will be followed immediately (within 10 min) after the breastfeeding session.

SUMMARY:
We aim to determine whether there are any differences in the UtA doppler measurements in postpartum women prior and right after breastfeeding.

DETAILED DESCRIPTION:
There is emerging evidence linking abnormal UtA Doppler indices in the postpartum period as a risk factor for developing future cardiovascular disorders. Thus far, no study considered the postpartum physiology itself as a possible confounder. If one wishes to draw conclusions about future cardiovascular risk, the role of oxytocin as a confounder must be determined. In the current study, we aim to determine whether oxytocin, physiologically produced during breastfeeding, has an effect on the UtA Doppler measurements in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

-Every woman who had vaginal delivery, instrumental delivery or cesarean section.

Exclusion Criteria:

-Patient's refusal, women who decided not to breastfeed, women who wish to breastfeed, but in whom no milk production commenced yet.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Postpartum women
Study Population: Every woman who had vaginal delivery, instrumental delivery or cesarean section.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum uterine artery doppler changes prior and after breastfeeding. | One year
  To determine whether there are any differences in the UtA doppler measurements in postpartum women prior and right after breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Yaniv Zipori, M.D, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided